CLINICAL TRIAL: NCT01882075
Title: Automated Administration of Fluid Administration Thanks to Hemodynamic Parameters and Cardiac Output During General Anesthesia
Brief Title: Closed-loop Fluid Administration System: Pilot Study to Evaluate Feasibility
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Dysfonction of the device
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/17; 2012-A00610-43 (Other: ANSM)
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia
Keywords: Anesthesia; Fluid administration; Closed-loop

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open loop (Active Comparator): fluid replacement (hydroxyethyl starch 130/0.4) is decided by the physicians according to continuous cardiac output measured by LidCO rapid device
  Interventions: Drug: Open loop
- Closed-loop (Experimental): Fluid replacement is automated. An algorithm has been developed ; the input value is continuous cardiac output measured by LidCO rapid device; the computer steers iv infusion of hydroxyethyl starch 130/0.4.
  Interventions: Device: Closed-loop

INTERVENTIONS:
Drug: Open loop
  Other Names: fluid replacement by Voluven(hydroxyethyl starch 130/0.4)
  Arms: Open loop
Device: Closed-loop
  Other Names: fluid replacement by Voluven (hydroxyethyl starch 130/0.4) is automated (closed-loop)
  Arms: Closed-loop

SUMMARY:
The investigators want to test during anesthesia the feasibility of a closed-loop automated fluid replacement system using cardiac output monitoring as the input value.

DETAILED DESCRIPTION:
The optimization of the cardiac output is an important goal during anesthesia to decrease the postoperative morbidity, mortality and the care costs.

We want to test if the closed-loop fluid administration is feasible.

Two groups will be compared. In all cases:

* anesthesia will be provided by a closed-loop which aim is to maintain bispectral index between 40 and 60 using propofol and remifentanil. This method permits to have similar depths of anesthesia in all cases.
* cardiac output will be continuously monitored by LidCO. In one group, fluid replacement is decided by the physician; in the other, fluid replacement is automated using a closed-loop system.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-75 years
* Scheduled for abdominal surgery under general anesthesia and requiring an invasive arterial blood pressure monitoring
* Consenting to participate in the study

Exclusion Criteria:

* Pregnant, breast feeding women
* Allergy
* Pacemaker
* Psychiatric disease, dementia, brain disease
* Contraindication to hydroxyethyl starch
* Inability to measure pulse pressure variability : arrhythmia, spontaneous breathing, or tidal volume < 7 ml/Kg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Mean cardiac output index during the surgery | One day after anesthesia

SECONDARY OUTCOMES:
Time before reaching maximizing cardiac output | One day after anesthesia
Volume of fluid replacement during surgery | One day after anesthesia
cardiac index during the surgery | One day after anesthesia
  Maximum and minimum values during the surgery
arterial hypertension | One day after anesthesia
  Number of events treated
Dysfunction of the closed-loop fluid device | One day after anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Foch, Suresnes, France